CLINICAL TRIAL: NCT00102453
Title: An Open-Label Pilot Study of Pentoxifylline in Steroid-naive Duchenne Muscular Dystrophy
Brief Title: Pentoxifylline in Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Responsible Party: CINRG Medical Director, CINRG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNMC0302
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Duchenne; Genetics
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Solution (Experimental): All enrolled participants were give pentoxifylline in this pilot protocol.
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline dosing: 20mg/Kg/day in a 20 mg/mL solution. Maximum dose of 1200mg/day. Dosing split into two equal parts taken morning and night with food.
  Other Names: Supplier: Frank's Pharmacy, Ocala, Fl. 34474.; Product: Pentoxifylline BP; CAS number: 5/6/6493; Formula weight: 278.35; Chemical formula: C13H18N4O3

SUMMARY:
In this study, the primary aim will be to estimate the magnitude and variability of strength change over time that may be expected for subjects on the study treatment. This estimate of effect will allow us to develop a rigorous statistical plan in the future randomized study. The specific estimation technique to be applied will use a linear random effects model to estimate average strength change during the 3-month lead-in period and then during the twelve-month treatment period, taking into account the quantitative muscle testing (QMT) measures for each subject. Accounting for the correlation between repeated measures from each subject by using a random effects model will yield an unbiased estimate of variability for the population average change in strength. We will use an analysis of pre- and post-treatment data to inform a best estimate of treatment effect. For example, the difference in QMT trends pre- and post-treatment would provide a straightforward measure of efficacy.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is a progressive disease of skeletal muscle caused by the absence of dystrophin due to a genetic mutation in the x-linked dystrophin gene. The absence of dystrophin results in a fragile muscle membrane that permits an abnormal permeability to electrolytes, especially Ca ++. The increase in intracellular calcium triggers a pathological cascade of events that ultimately results in muscle necrosis and fibrosis, which impedes normal muscle regeneration. The increased knowledge of the pathophysiology of DMD opens the opportunity for pharmacological treatment, with the purpose of altering the disease process and or reverting the muscle degeneration.

This research study requires having Duchenne muscular dystrophy (DMD) and the subject to be between 4 and 7 years old. We expect 5 children to take part in this study at Children's Hospital and 10 other children to participate at other hospitals worldwide.

There will be two (2) screening visits to help decide whether you will be able to participate in the study. At the second screening visit, there will be a blood test (about 13 tablespoons of blood), and an EKG. Once the study doctors decide eligibility to be in the study, the subject will then come back once a month for three months to have his strength tested. After three months, the subject will begin to take the pentoxifylline and have an MRI (you will have a test called an MRI to look inside the muscles of your legs). This will continue for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age 4 to 7 years
3. Ambulant independently. Subjects may use a wheelchair occasionally, but only for long distances
4. Diagnosis of DMD confirmed by at least one of the following:

   * Dystrophin immunofluorescence and/or immunoblot showing complete dystrophin deficiency, and clinical picture consistent with typical DMD OR
   * Gene deletion test positive (missing one or more exons) in the central rod domain (exons 25-60) of dystrophin, where reading frame can be predicted as 'out-of-frame',
   * and clinical picture consistent with typical DMD.
   * Complete dystrophin gene sequencing showing an alteration (point mutation, duplication, or other mutation resulting in a stop codon mutation) that can be definitely associated with DMD, with a typical clinical picture of DMD.
5. Positive family history of DMD confirmed by one of the criteria listed above in a sibling or maternal uncle, and clinical picture typical of DMD.
6. Glucocorticosteroid - naïve (i.e. has not been treated with prednisone or Deflazacort within 1 year before onset of the study)
7. Has not participated in other therapeutic research protocol within the last 6 months.
8. Evidence of muscle weakness by MRC score or clinical functional evaluation
9. Ability to provide reproducible repeat QMT bicep score of either the right or left arm within 15% of first assessment score.

Exclusion Criteria:

1. Symptomatic DMD carrier
2. Use of any medication, nutritional supplement or herb for treatment of DMD within the last 3 months.
3. Symptomatic cardiomyopathy or ventricular arrhythmias
4. History of significant concomitant illness, impairment of blood clotting ability (as evidenced by increased PT/PTT or bleeding time over the upper limit of normal (ULN)), recent cerebral or retinal hemorrhage, bleeding diathesis, gastric ulcer, hypotension or significant impairment of renal or hepatic function (defined as serum creatinine and GGT respectively, greater than 1.5 times normal upper limit for age and gender).

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2002-03; Primary Completion 2006-07 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
QMT measurements | Each study visit
  Quantitative muscle testing (QMT) is a technique utilized to assess muscle strength. Measurements of force are collected using a load cell while performing a maximum voluntary isometric contraction. This set-up is able to measure changes in strength of 0.25 lb which provides accurate and sensitive measurement of muscular strength. QMT is performed by a CINRG physical therapist.

SECONDARY OUTCOMES:
Change in manual muscle test (MMT) at 12 months | Each study visit
  Manual muscle testing (MMT), which is graded according to the modified Medical Research Council (MRC) scale, is a test of a participant's muscle strength, or ability of the muscle to move a part of the body against resistance. A CINRG physical therapist will perform MMT testing with each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Escolar, MD, Study Chair — Children's National Research Institute
Locations (5):
- United States (5):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic, Rochester, Minnesota
  - Washington University at St. Louis, St Louis, Missouri
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Scottish Rite Hospital, Dallas, Texas